CLINICAL TRIAL: NCT02208050
Title: A Phase IV Double Blind, Randomized, Placebo Controlled, Crossover Study of the Effectiveness of Oral Fampridine in Improving Upper Limb Function in Progressive Multiple Sclerosis
Brief Title: A Study of the Effectiveness of Fampridine in Improving Upper Limb Function in MS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University College Dublin (Other)
Responsible Party: Principal Investigator, Christopher McGuigan, Consultant Neurologist, University College Dublin
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SVUHneuro002
Record Dates: First submitted 2014-05-19; First posted 2014-08-04 (Estimated); Results first posted 2021-07-09 (Actual); Last update posted 2021-07-09 (Actual); Status verified 2021-07

CONDITIONS: Secondary Progressive Multiple Sclerosis; Primary Progressive Multiple Sclerosis
Keywords: Secondary Progressive Multiple Sclerosis; Primary Progressive Multiple Sclerosis; Multiple Sclerosis; Upper limb function; Mobility; Fampridine; DASH; AMSQ; MSWS-12; MSIS-29; SF-36; 9HPT; 25FTW; JTT
MeSH Terms: conditions — Multiple Sclerosis, Chronic Progressive; Multiple Sclerosis | interventions — 4-Aminopyridine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 1 (Other): Patients will be randomised to a 8 week treatment period with the active drug followed by a 2 week washout period before an 8 week treatment period with placebo.
  Interventions: Drug: Fampridine; Drug: Placebo
- Group 2 (Other): Patients will be randomised to a 8 week treatment period with the placebo, followed by a 2 week washout period and a further 8 week treatment period with the active drug.
  Interventions: Drug: Fampridine; Drug: Placebo

INTERVENTIONS:
Drug: Fampridine
  Other Names: Fampyra
Drug: Placebo

SUMMARY:
The purpose of this study is to examine the effect of treatment with fampridine in patients with secondary progressive MS (SPMS) or primary progressive MS (PPMS) with upper limb dysfunction (as defined by a 9-HPT time of between 15-90 seconds) and Kurtzke EDSS scores in the range 4.0-7.0 on upper limb function assessed by the nine-hole peg test (9-HPT) and the Jebson Taylor Hand Function Test (JTT).

Fampridine has been shown to be effective in improving motor function, specifically walking ability in prior studies in this patient population and is currently licensed for this use in Europe and the United States. Upper limb dysfunction is common in SPMS and PPMS and often underestimated. Fampridine effects action potential conduction in demyelinated nerve fibres and we would hypothesise that the improvement previously reported in walking ability would be similar to that on upper limb dysfunction. Our study aims to address this question using both independent and patient reported outcomes in the context of a randomised placebo controlled crossover trial.

DETAILED DESCRIPTION:
BACKGROUND INFORMATION Patients with secondary progressive MS (SPMS) and primary progressive MS (PPMS) have significant walking disability and impaired upper limb function due to repeated demyelination and axonal injury affecting the corticospinal pathways. In some patients this motor deficit may be predominantly due to demyelination resulting in motor conduction slowing and/or block which is potentially reversible by blocking potassium channels of demyelinated axons. Fampyra® (fampridine-PR) is a prolonged-release formulation of the active drug substance 4-aminopyridine {4-AP; fampridine [International Nonproprietary Name (INN)]. Fampridine is able to block certain voltage-gated K+ channels in neurons, particularly in demyelinated nerves. Blockade of repolarising K+ currents can increase synaptic transmission throughout the nervous system by increasing the duration of the presynaptic action potential. Demyelinated nerves lose their ability to effectively conduct action potentials and fampridine can help reverse this. This effect was demonstrated clinically in a proportion of multiple sclerosis (MS) patients who showed a significant improvement in motor function, specifically walking ability, with Fampyra treatment. Fampridine-PR 10 mg every 12 hours or twice daily (BID) was approved in Europe (20 July 2011) for this indication under the brand name of Fampyra®.

RATIONALE FOR THE STUDY Treatment with fampridine (4-aminopyridine), a potassium channel blocker,1,2 has been shown to cause significant improvement in walking speed in one third of MS patients with motor disability.3-5 In those patients who respond, approximately a 25% improvement in walking speed was obtained with a self-reported 7 point improvement in the Multiple Sclerosis Walking Scale (MSWS-12), a patient-rated measure of walking quality and ability, 6,7 in comparison to non-responding patients and placebo control subjects.

Pharmacologically, the K+ channel blocking properties of fampridine and its effects on action potential conduction in demyelinated nerve fiber preparations have been extensively characterized. At low concentrations that are relevant to clinical experience (in the range of 0.2 to 2 μM [18 to 180 ng/mL]), fampridine is able to block certain voltage-dependent K+ channels in neurons. It is this characteristic that appears to explain the ability of the drug to restore conduction of action potentials in some critically demyelinated nerve fibers. At higher (millimolar) concentrations, fampridine affects other types of K+ channels in both neural and non-neural tissues. Blockade of repolarising K+ currents may increase synaptic transmission throughout the nervous system by increasing the duration of the presynaptic action potential. A range of neurological effects consistent with increased excitability of nerve cells occurs with clinically relevant doses of fampridine.

The FDA has recently approved Fampridine, a slow release preparation, for use in the MS patient population.8 It has also recently been approved in Europe (20th July 2011).17 Most studies of fampridine assessed timed walking over twenty-five feet and the Multiple Sclerosis Walking Scale-12 (MSWS-12).3-5 Deficits in arm and hand function are commonly found in patients with SPMS and PPMS and can have an impact in performing many activities of daily living. We propose to examine the efficacy of fampridine in upper limb function and in overall disease impact in a single centre, double blind, randomized, placebo-controlled, crossover study of patients attending St Vincent's University Hospital with significant walking and upper limb disability due to SPMS and PPMS.

STUDY OBJECTIVE

The objective of this study is to assess the affect of PR-fampridine medication compared to placebo for upper limb function in patients with progressive multiple sclerosis

TRIAL DESIGN

This will be a single centre, phase IV, double blind, randomized, placebo controlled, crossover study on the effectiveness of oral Fampridine-PR 10mg tablets BID on upper limb function for patients with progressive multiple sclerosis.

The trial will consist of a two week run in period followed by an eight week treatment period were enrolled subjects will be randomised to receive either study drug or placebo in a double blinded manner. This will be followed by a two-week wash out period followed by a further eight-week study period using active drug or placebo. There will be a two-week washout period at the end of the study. The total period of the study will be 22 weeks.

Each subject will attend for a screening visit and 8 assessment visits (total number of visits, 9).

STUDY ASSESSMENTS AND PROCEDURES

Patients likely to fulfill the inclusion criteria and not meet any exclusion criteria will be provided with information on the study and invited to attend a subsequent screening visit. Only patients who have signed the informed consent form will participate in any study related procedures including blood testing and ECG.

At screening visit (Assessment 1) subjects will have a physical examination and an expanded disability status scale (EDSS) score rated. Blood samples will be taken for renal and liver function and a baseline ECG performed. Patients will complete a nine-hole peg test (9-HPT) and a Jebsen Taylor Hand Function Test (JTT). Timed 25 foot walk (T25FW) will be recorded and the patients invited to complete the Multiple Sclerosis Impact Scale (MSIS-29), Multiple Sclerosis Walking Scale (MSWS-12), Disabilities of the Arm, Shoulder and Hand (DASH) score, Arm Function in Multiple Sclerosis Questionnaire (AMSQ) and SF-36 (quality of life) questionnaire. Patients with any abnormalities on ECG, blood tests will not be invited to a baseline visit and considered a screening failure.

Following screening visit subjects fulfilling the inclusion / exclusion criteria will have two baseline visits (Assessments 2 and 3) at the end of week one and end of week two. The 9-HPT, JTT and T25FW will be repeated to allow for training effects. Patients will be randomised to group A or group B and receive study medication or placebo at baseline visit based on their blinded randomisation (Assessment 3).

The first treatment period will be from the start of week 3 until the end of week 10. Patients will have an assessment at the end of week 6 (Assessment 4) and the end of week 10 (Assessment 5). At both assessments patients will have the 9-HPT, JTT, T25FW, MSIs-29, MSWS-12, DASH, AMSQ and SF-36 recorded. Weeks 11 and 12 will be a washout period (no drug/placebo). Assessment 6 will occur at the end of week 12 and will include recording of 9-HPT, JTT, T25FW, MSIs-29, MSWS-12, DASH, AMSQ and SF-36. Any adverse events will be recorded at each visit as will the use of concomitant medications.

The second treatment period will begin at the start of week thirteen with groups A and B switching study drug / placebo in a blinded manner. The second treatment period will continue for a further 8 weeks with two more assessments ant week 16 (Assessment 7) and week 20 (Assessment 8). At both of these assessments subjects will complete the 9-HPT, JTT, T25FW, MSIs-29, MSWS-12, DASH, AMSQ and SF-36. At the end of week 20 and EDSS score will be recorded. Any adverse events will be recorded at each visit as will the use of concomitant medications.

There will be a final washout period (weeks 21 and 22) after which a final visit (assessment 9) will occur and subjects once again completing 9-HPT, JTT, T25FW, MSIS-29, MSWS-12, DASH, AMSQ and SF-36 and having n EDSS score recorded. Once again adverse events will be recorded.

Description of Study Assessments

Medical and Surgical History will be recorded with particular attention on the diagnosis of MS, duration of MS and MS subtype.

Demographics The date of birth, gender and race will be recorded. Physical Examination The complete physical examination will include the evaluation of the neurological system and a recording of the EDSS score and T25FW.

ECG Test One ECG including a 12-lead examination will be performed at Screening (assessment 1).

Abnormal findings will be noted for clinical significance. The report will be signed by the investigator.

Clinical Laboratory Tests

1. Haematology: haemoglobin, WBC, RBC, platelet count
2. Biochemistry: creatinine or creatinine-clearance, sodium, potassium, liver function tests
3. All laboratory results will be reviewed and the reports signed by the investigator who will record in the CRF whether they are normal, abnormal but not clinically significant, or abnormal and clinically significant.

Pregnancy Tests Serum pregnancy test and urine pregnancy test in women of childbearing potential will be performed.

Concomitant Medication In addition to Fampyra, any other treatments or procedures that are considered necessary for the patient's welfare may be given at the discretion of the Investigator. Administration of continuous concomitant procedures and medications (including herbals and nutraceuticals) must be reported in the appropriate section of the CRF along with reasons for use. Continuous concomitant procedures and medications are defined as a treatment administered regularly for 2 weeks or more. The generic names for concomitant medications should be recorded, if possible. The total daily dose should be recorded in the CRF whenever possible. Concomitant use of medicinal products that are inhibitors of OCT2 for example, cimetidine will be noted and will be deemed exclusion criteria. Concomitant use medicinal products that are substrates of OCT2 for example, carvedilol, propanolol and metformin will also be noted and the investigator will decide if the subject should successfully complete screening.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be able and willing to give written informed consent and to comply with the requirements of this study protocol
* Subjects must be diagnosed with clinically definite SPMS or PPMS and be judged to be in generally good health by the investigator based upon the results of the medical history, laboratory tests (liver and renal function), physical examination, 12-lead electrocardiogram performed during Screening
* Subjects must be Male or female aged 18-70 at baseline
* Kurtzke EDSS scores in the range 4.0 to 7.0 inclusive
* Evidence of significant upper limb dysfunction as defined by a 9HPT of 15 - 90 seconds (dominant or non-dominant hand)
* Female subjects with reproductive capabilities must have a negative serum pregnancy test at baseline and agree to using an acceptable form of contraception for the duration of the study (barrier, coil or oral contraceptives only).

Exclusion Criteria:

* Allergy/sensitivity to study medications or their ingredients
* Female subjects who are pregnant or breast-feeding or considering becoming pregnant during the study.
* Subjects unable to provide written informed consent
* Subjects with a history of epilepsy or previous seizures (including provoked seizures).
* Subjects who have a history of drug or alcohol use that, in the opinion of the investigator, would interfere with adherence to study requirements.
* Subjects with an AST or ALT ≥ 3 x ULN on liver function tests
* Subjects have clinically significant ECG findings as judged by the investigator, in particular evidence of a cardiac conduction defect.
* Significant upper or lower limb arthritis as considered by the investigator to interfere with study assessments.
* Significant cognitive impairment as considered by the investigator to interfere with study assessments
* Subjects with clinically significant upper limb ataxia considered by the investigator to interfere with ability to complete study outcome measures.
* Patients with mild, moderate or severe renal impairment (creatinine clearance<80ml/min) measured by 24-hour urine collection or estimated by the Cockcroft and Gault formula
* Subjects concomitantly using medicinal products that are inhibitors of Organic Cation Transporter 2 (OCT2) for example cimetidine
* Concurrent treatment with other medicinal products containing fampridine (4- aminopyridine)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2014-02-21 (Actual); Primary Completion 2016-02-16 (Actual); Study Completion 2016-02-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher McGuigan, MD, Principal Investigator — University College Dublin, St Vincent's University Hospital
Locations (2):
- Ireland (2):
  - St Vincent's University Hospital, Dublin, Dublin 4
  - St. Vincents University Hospital, Dublin

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study recruited male and female patients between the ages of 18 - 70 years with clinically definite primary or secondary progressive multiple sclerosis, between 2013 and 2015. After recruitment and randomisation, three baseline assessments occurred over two weeks. Patients were then treated with fampridine-washout-placebo or placebo-washout-fampridine for 8 weeks followed by a 2 week washout and then cross-over to the other arm for 8 weeks followed by a 2 week washout.
Groups:
- Group A: Fampridine Followed by Placebo: Participants who received fampridine first before crossing over to the placebo arm. Following baseline assessment and randomisation, participants received 10mg pr-fampridine twice daily for eight weeks followed by a two week washout period and then received placebo tablet twice daily for ten weeks.
- Group B: Placebo Followed by Fampridine: Participants who received placebo first before crossing over to fampridine. After baseline assessment and randomisation, participants received placebo twice daily for 8 weeks, then had a 2 week washout period, followed by 8 weeks of treatment with 10mg pr-fampridine.
Period: Baseline Assessment Period: 2 Weeks
Arm/Group | Group A: Fampridine Followed by Placebo | Group B: Placebo Followed by Fampridine
Started | 36 | 28
Completed | 36 | 28
Not Completed | 0 | 0
Period: Treatment Period 1: 8 Weeks Treatment
Arm/Group | Group A: Fampridine Followed by Placebo | Group B: Placebo Followed by Fampridine
Started | 36 | 28
Completed | 36 | 28
Not Completed | 0 | 0
Period: Washout Period 1: 2 Weeks
Arm/Group | Group A: Fampridine Followed by Placebo | Group B: Placebo Followed by Fampridine
Started | 36 | 28
Completed | 35 | 28
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0
Period: Treatment Period 2: 8 Weeks Treatment
Arm/Group | Group A: Fampridine Followed by Placebo | Group B: Placebo Followed by Fampridine
Started | 35 | 28
Completed | 33 | 28
Not Completed | 2 | 0
Period: Washout Period 2: 2 Weeks Washout.
Arm/Group | Group A: Fampridine Followed by Placebo | Group B: Placebo Followed by Fampridine
Started | 33 | 28
Completed | 33 | 28
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Group 1: Fampridine Followed by Placebo: Patients will be randomised to a 8 week treatment period with the active drug followed by a 2 week washout period before an 8 week treatment period with placebo.
  Fampridine
  Placebo
- Group 2: Placebo Followed by Fampridine: Patients will be randomised to a 8 week treatment period with the placebo, followed by a 2 week washout period and a further 8 week treatment period with the active drug.
  Fampridine
  Placebo
- Total: Total of all reporting groups
Arm/Group | Group 1: Fampridine Followed by Placebo | Group 2: Placebo Followed by Fampridine | Total
Number analyzed (Participants) | 36 | 28 | 64
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 33 | 25 | 58
  >=65 years | 3 | 3 | 6
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 55.1 [45.1 to 59.5] | 53.7 [45.4 to 60.9] | 55.1 [45.4 to 60.2]
Sex: Female, Male [Count of Participants; unit: Participants]
  Sex: Female | 23 | 15 | 38
  Sex: Male | 13 | 13 | 26
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Ireland | 36 | 28 | 64
Multiple Sclerosis (MS) Subtype [Count of Participants; unit: Participants]
  Secondary Progressive MS (SPMS) | 23 | 22 | 45
  Primary Progressive MS (PPMS) | 13 | 5 | 18
  Unknown | 0 | 1 | 1
On Disease Modifying Treatment (DMT) [Count of Participants; unit: Participants] — Participants who are currently being treated with a licensed disease modifying treatment (DMT) (not including symptomatic treatments) for multiple sclerosis including Interferons and Glatiramer Acetate.
  Participants | 12 | 13 | 25
EDSS (Expanded Disability Status Scale) [Median (Full Range); unit: units on a scale] — Expanded Disability Status Scale is a measure designed to assess level of physical disability in multiple sclerosis, ranging from 0 - no detectable disability to 10 - death due to MS. Higher scores indicate higher levels of disability. Score of 6 indicates unilateral assistance required to mobilise, 6.5 indicates bilateral assistance required; 7 indicates predominantly using wheelchair.
  units on a scale | 6 [4 to 7] | 6 [4 to 7] | 6 [4 to 7]
Disease Duration [Median (Inter-Quartile Range); unit: years] | 15.7 [9.9 to 24.6] | 19.2 [9.0 to 25.4] | 16.8 [9.3 to 25.0]
Baclofen [Number; unit: participants] | 4 | 4 | 8
Tizanadine [Count of Participants; unit: Participants] | 3 | 1 | 4
Benzodiazepine [Count of Participants; unit: Participants] | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Classified as Upper Limb Responders on the 9 Hole Peg Test (9HPT)
Description: 9 Hole Peg Test is a test of upper limb function. Participants place 9 pegs on pegboard and remove pegs - this is timed for each hand. Time recorded in seconds. Longer time indicates poorer upper limb function. 20% improvement is defined as 20% shorter time in seconds. An upper limb responder is defined as a patient with both of the two "on treatment" 9 Hole Peg Test (9-HPT) assessments measured in seconds (assessments 4 & 5 or 7 & 8) improving 20% from the average of the baseline assessments (1, 2 & 3). Washout assessment not included in the analysis.
Time Frame: 20 weeks. Baseline assessments 1,2,3: weeks 0-2. Assessment 4 - midway through first treatment period; assessment 5: end of first treatment period. Assessment 7: midway through second treatment period, assessment 8: end of second treatment period.
Population: Analysis population included all participants who received treatment and placebo for eight weeks. Two participants withdrew during the second 8-week treatment period and were not included in the final analysis.
Measure: Count of Participants; unit: Participants
Groups:
- PR-Fampridine: 10mg fampridine twice daily for 8 weeks.
- Placebo: Placebo tablets twice daily for 8 weeks.
Arm/Group | PR-Fampridine | Placebo
Number analyzed (Participants) | 62 | 62
Participants
  Dominant hand: Responders | 4 | 3
  Dominant hand: Non-responders | 58 | 59
  Non-dominant hand: Responders | 2 | 1
  Non-dominant hand: Non-responders | 60 | 61

2. Secondary Outcome: Number of Participants Defined as Upper Limb Responders on the Jebsen Taylor Hand Function Test (JTT)
Description: Jebsen Taylor Hand Function Test (JTT) is a timed test (seconds) comprising of seven 'real-world' tasks such as picking up small items. It has been validated for use in upper limb function in MS. A secondary measure of upper limb responsiveness will be defined as number of participants with a 20% improvement in from baseline in the average time taken to complete all seven tasks on the Jebsen Taylor Hand Function Test "on treatment" (assessments 4 & 5 or 7 & 8) compared with baseline assessments (assessments 1,2 & 3).
  Baseline assessments (1,2,3) performed in two week period prior to first treatment block. Longer time indicates worse functioning. Improvement is defined as shorter time in seconds.
  Assessment 4: Midway through first treatment period (week 4 of 8 week treatment period) Assessment 5: End of first treatment period (end of week 8) Assessment 7: Midway through second treatment period Assessment 8: End of second treatment period
Time Frame: 20 weeks: Weeks 0-2: Assessment 1/2/3; Week 6: Assessment 4; Week 10: Assessment 5; Week 16: Assessment 7; Week 20: Assessment 8
Population: Participants who had completed assessments at the above time points to allow analysis.
Measure: Count of Participants; unit: Participants
Groups:
- Fampridine: Fampridine 10mg bd treated participants in either Period 2 or Period 4.
- Placebo: Placebo treated participants in Period 2 and Period 4.
Arm/Group | Fampridine | Placebo
Number analyzed (Participants) | 63 | 61
Participants
  Dominant hand: Responders | 3 | 0
  Dominant hand: Non-responders | 60 | 61
  Non-dominant hand: Responders | 3 | 0
  Non-dominant hand: Non-responders | 60 | 61

3. Secondary Outcome: The Number of Mobility Responders to Fampridine as Measured by an Improvement in the 25 Foot Timed Walk (T25FW)
Description: A mobility responder to Fampridine will be defined as a patient with both of the two "on treatment" T25FW assessments (assessments 4 & 5 or 7 & 8) being better (shorter time in seconds) than the maximum of any of the four "off treatment" assessments (assessments 1, 2, 3, 6). Otherwise the patient will be deemed a non-responder. T25FW test is the time taken to walk 25 feet taken as the average of two trials. Measured in seconds. Longer time indicates slower walking. Improvement is considered shorter amount of time in seconds - no specific percentage or amount of time was considered necessary.
  Assessment 4: Midway through first treatment period (week 4 of 8 week treatment period) Assessment 5: End of first treatment period (end of week 8) Assessment 7: Midway through second treatment period Assessment 8: End of second treatment period.
Time Frame: as for outcome 2
Population: Population with 25 foot walk data on analysis of results.
Measure: Count of Participants; unit: Participants
Groups:
- Fampridine: Fampridine 10mg BD for eight weeks with baseline assessment and washout period.
- Placebo: Placebo BD for eight weeks with baseline assessment and washout period.
Arm/Group | Fampridine | Placebo
Number analyzed (Participants) | 61 | 61
Participants
  Responders | 59 | 59
  Non-responders | 2 | 2

4. Secondary Outcome: Mean Scores in DASH - Fampridine and Placebo.
Description: Disabilities of the Arm Shoulder and Hand Scores questionnaire: The DASH consists of a 30-item disability symptom scale scored 0 (no disability) to 100, developed as a self-rated upper extremity disability and symptoms. Higher scores indicate higher self-perception of disability.
  DASH questionnaire administered to fampridine treated group at Weeks 6,10,16 and 20. Scores at each time point were summed and averaged. DASH questionnaire administered to placebo treated group at Weeks 6,10,16 and 20. Scores at each time point were summed and averaged.
Time Frame: 20 weeks: Assessments at Week 6 - midway through first treatment period, Week 10 - end of first treatment period, Week 16 - midway through second treatment period, Week 20 - end of second treatment period.
Population: Mean scores in the DASH for all participants in the trial during on treatment periods (assessments 4&5; 7&8).
Measure: Mean (Standard Deviation); unit: Mean units on a scale.
Groups:
- Fampridine: Average scores for participants treated with fampridine during weeks 2-10 or weeks 12-20.
- Placebo: Average scores for patients when treated with placebo during weeks 2-10 or weeks 12-20.
Arm/Group | Fampridine | Placebo
Number analyzed (Participants) | 63 | 63
Mean units on a scale. | 35.4 (19.5) | 38.3 (20.5)

5. Secondary Outcome: Mean Scores in Multiple Sclerosis Walking Scale (MSWS-12) - Fampridine and Placebo.
Description: Multiple Sclerosis Walking Scale 12 is a 12-item self report measure of the impact of MS on an individual's walking ability. Scores are summed 1-3; 1-5 for each item. Higher scores indicate higher limitation in walking ability. Scores are summed and transformed to a 0-100 scale again with higher scores indicating higher self-reported limitation in walking ability. MSWS12 scores were collected for the group on Placebo treatment at Weeks 6,10,16 and 20 - the sum of the 4 scores was averaged. MSWS-12 scores were collected for the group on Fampridine treatment at Weeks 6, 10, 16, 20. The sum of the 4 scores was averaged.
Time Frame: as for outcome 4
Population: Participants on treatment with Fampridine or Placebo.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- On Treatment: Fampridine: Assessments during on-treatment periods with fampridine.
- Placebo: Assessments during on-treatment periods with Placebo.
Arm/Group | On Treatment: Fampridine | Placebo
Number analyzed (Participants) | 62 | 62
units on a scale | 64.5 (28.2) | 65 (27)

6. Secondary Outcome: Mean Scores in the Disabilities in Arm Function in Multiple Sclerosis Questionnaire (AMSQ) Score Between Fampridine and Placebo.
Description: AMSQ - Arm Function in Multiple Sclerosis Questionnaire. This is a 31-item patient reported outcome measure which is validated to measure limitation in arm and hand functioning in people with multiple sclerosis. Patients rate the ability to which they can perform routine daily tasks with current hand function. Higher scores indicate greater limitations. Scale ranges from 0-100. AMSQ scores were collected for the group on Placebo treatment at Weeks 6,10,16 and 20 - the sum of the 4 scores was averaged. AMSQ scores were collected for the group on Fampridine treatment at Weeks 6, 10, 16, 20. The sum of the 4 scores was averaged.
Time Frame: as for outcome 4
Population: Mean scores on AMSQ during on-treatment period. (AMSQ assessments 4 & 5, 7 & 8).
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Fampridine: Assessments while participants on treatment with fampridine (4&5 or 7&8).
- Placebo: Assessments while on treatment with placebo (4&5 or 7&8)
Arm/Group | Fampridine | Placebo
Number analyzed (Participants) | 62 | 62
units on a scale | 35.4 (19.8) | 38.4 (21.5)

7. Secondary Outcome: Mean Scores of MSIS-29 - Fampridine and Placebo
Description: MSIS-29 is a patient reported outcome with a physical and psychological component combined into one scale. They refer to the self-reported impact of MS on their physical and psychological wellbeing. Higher scores indicate a higher impact on functioning. The 20 item physical scale and the 9 item psychological scale are reported as two separate scaled scores. Both scale ranges are 0-100. Higher scores indicate a higher impact on functioning. MSIS -20 and MSIS-9 scores were collected for the group on Placebo treatment at Weeks 6,10,16 and 20 - the sum of the scores was averaged. MMSIS-20 and MSIS-9 scores were collected for the group on Fampridine treatment at Weeks 6, 10, 16, 20. The sum of the scores was averaged.
Time Frame: as for outcome 4
Population: Participants during on-treatment period with fampridine or placebo.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Fampridine: MSIS-20: MSIS-20 scores during treatment with fampridine.
- Placebo: MSIS20: MSIS-20 scores during treatment with placebo.
- Fampridine: MSIS-9: MSIS-9 scores during treatment with fampridine
- Placebo: MSIS-9: MSIS-9 scores during treatment with placebo.
Arm/Group | Fampridine: MSIS-20 | Placebo: MSIS20 | Fampridine: MSIS-9 | Placebo: MSIS-9
Number analyzed (Participants) | 62 | 62 | 62 | 62
units on a scale | 42.4 (22) | 43.3 (24) | 30.5 (22) | 29.4 (21)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected for each participant for the study period (22 weeks).
Groups:
- Fampridine: Adverse events reported by the patients when treated with Fampridine
- Placebo: Adverse events reported by the patients when treated with placebo.
Arm/Group | Fampridine | Placebo
All-Cause Mortality (participants affected / at risk) | 0/64 | 0/64
Serious Adverse Events (participants affected / at risk) | 0/64 | 0/64
Other Adverse Events (participants affected / at risk) | 32/64 | 25/64
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fampridine (N=64) | Placebo (N=64)
Peripheral venous disease (Vascular disorders) | 1 (1) | 0 (0)
Laceration to Foot (Injury, poisoning and procedural complications) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 2
Elevated hepatic enzymes (Investigations) | 3 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Lymphopenia (Blood and lymphatic system disorders) | 1 | 2
Thrombocytosis (Blood and lymphatic system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 5 | 4
Headache (Nervous system disorders) | 7 | 0
Worsening hemiparesis (Nervous system disorders) | 2 | 1
Muscle Spasticity (Nervous system disorders) | 2 | 0
Numbness (Nervous system disorders) | 0 | 2
Tremor (Nervous system disorders) | 2 | 1
Syncope (Nervous system disorders) | 3 | 0
Influenza like illness (General disorders) | 1 | 0
Fatigue (General disorders) | 3 | 1
Insomnia (General disorders) | 1 | 1
Weakness (General disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 4 | 0
Vomiting (Gastrointestinal disorders) | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 1
Constipation (Gastrointestinal disorders) | 0 | 2
Rash (Skin and subcutaneous tissue disorders) | 0 | 1
Mobility (Musculoskeletal and connective tissue disorders) | 1 | 3
Muscular pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Pain extremity (Musculoskeletal and connective tissue disorders) | 2 | 3
Hip Pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0
Ear Infection (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 1 | 0
Urinary Tract Infection (Infections and infestations) | 2 | 3
Sinusitis (Infections and infestations) | 1 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 5 | 0
Lower Respiratory Tract Infection (Infections and infestations) | 2 | 1
Influenza (Infections and infestations) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2013-02-03): https://cdn.clinicaltrials.gov/large-docs/50/NCT02208050/Prot_SAP_000.pdf